CLINICAL TRIAL: NCT04993872
Title: Pharmacokinetics of Calcineurin & mTOR Inhibitors in HIV-1 Infected Kidney Transplant Recipients After Switch to BIC/FTC/TAF: a Pilot Study - KINETIK (KIdNEy Transplant bIKtarvy) IMEA 064
Brief Title: Pharmacokinetics of Calcineurin & mTOR Inhibitors in HIV-1 Infected Kidney Transplant Recipients After Switch to BIC/FTC/TAF
Acronym: KINETIK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: INSERM UMR S 1136 (Other); Sebastien GALLIEN/Henri Mondor University Hospital- Infectiology Department (Unknown); THOMAS STEHL/ HENRI MONDOR HOSPITAL-Department of Nephrology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 064
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2022-10

CONDITIONS: HIV-infected Patient Kidney Transplant Recipient
Keywords: HIV+,,KIDNEY TRANSPLANT, BIKTARVY,cALCINEURIN? mTOR
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIC/FTC/TAF (Experimental): Development phase 4: Biktarvy®
  Interventions: Drug: Biktarvy Tab

INTERVENTIONS:
Drug: Biktarvy Tab — Multicenter Pilot study aiming to assess the safe use of BIC/FTC/TAF in HIV-KTR, using a single-arm design.

SUMMARY:
Chronic kidney disease (CKD) is a critical comorbidity for patients living with HIV (PLWH), with an estimated prevalence between 2.4 and 17%, leading to end-stage renal disease 3 to 6 fold more than non-HIV population. However kidney transplantation for PLWH has become the first-line therapy for end-stage renal disease, with an enhanced survival benefit compared to remaining on dialysis.

Management of antiretroviral therapy (ART) in HIV-infected kidney transplant recipients (HIV-KTR) has historically been problematic because of the potential nephrotoxicity of some antiretroviral drugs and the interactions between calcineurin inhibitors, mTOR inhibitors, and ritonavir or cobicistat-boosted containing-ART. The use of tenofovir disoproxil fumarate (TDF), a widely recommended nucleotide analogue for the treatment of both HIV and HIV/hepatitis B virus (HBV) co-infection, is restricted in vulnerable kidney population as HIV-KTR due to its major potential toxicity consistent with tubular dysfunction and rarely with a progressive sustained decline in renal function. The optimal long-term ART regimen is not known in HIV-KTR, though it makes intuitive sense to avoid regimens containing TDF, given its potential nephrotoxicity. Nevertheless the potent virological efficacy of TDF both on HIV and HBV and its highest in-vitro barrier to resistance among the Nucleoside Reverse Transcriptase Inhibitors makes tenofovir use highly recommended or even essential in HIV/HBV co-infections.

Tenofovir alafenamide (TAF) and bictegravir (BIC) are 2 novel antiretroviral drug available in HIV treatment in combination with emtricitabine (F) (B/F/TAF):

* TAF is a novel prodrug of tenofovir that may offer improved renal safety over TDF. TAF is more stable in plasma and is metabolized intracellularly by cathepsin A, an enzyme that is highly expressed in lymphoid tissues. Therefore, TAF can achieve higher intracellular levels of the active moiety tenofovir diphosphate, with lower levels of circulating tenofovir when compared with TDF. This more targeted treatment could potentially result in fewer renal and bone complications despite the same clinical efficacy as TDF. TAF was approved for use in PLWH with mild-moderate CKD (eGFR: 30-69 mL/min).

The availability of TAF seems a potential addition to the antiretroviral armamentarium in HIV-KTR. * BIC is a novel second-generation integrase strand transfer inhibitor (INSTI) has a high in-vitro barrier to resistance and in-vitro activity against most INSTI-resistant variants and has low potential for clinically meaningful drug-drug interactions. BIC has been recently approved by the FDA, in coformulated B/F/TAF for the treatment of HIV-1 infection in antiretroviral naïve subjects and in those with suppressed viremia.

No data are available yet with TAF use in HIV-infected kidney transplant recipients as well as with BIC, especially about potential drug-to-drug interactions with immunosuppressive drugs such as calcineurin & mTOR inhibitors.

At last simplification to a single tablet regimen (STR) may offer a once-daily option for HIV-KTR who have multiple comorbidities, often requires complex regimens with a high pill burden.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients > 18 years
* Kidney transplant recipient ≥ 3 months
* Receiving calcineurin and/or mTOR inhibitors without change in doses ≥ 4 weeks
* Plasma HIV RNA ≤ 50 cpml ≥ 6 months (1 blip permitted <200cp/ml)
* eGFR (CKD-EPI) ≥ 30 ml/mn/1.73m2
* Written consent
* GSS to BIC/FTC/TAF GSS ≥ 2
* stable antiretroviral regimen for at least 3 months
* Active contraception in potential child-bearing women

Exclusion Criteria:

* Allergy or intolerance to one of the following drug or to any of excipients: FTC, TDF, INSTI
* HIV-2 or HIV-1/HIV-2 co-infection
* Patients with severe hepatic impairment (Child-Pugh Class C)
* Patient without health coverage
* Pregnancy and breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in calcineurin & mTOR inhibitors' blood concentrations after switch to B/F/TAF | Week 2
  Evolution of blood concentration

SECONDARY OUTCOMES:
•Proportion in calcineurin & mTOR inhibitors' dose changes after switch to B/F/TAF | Baseline
  PK of calcineurin and mTOR
•Proportion in calcineurin & mTOR inhibitors' dose changes after switch to B/F/TAF | Week 2
  PK of calcineurin and mTOR
• Changes in plasma levels of calcineurin & mTOR inhibitors | Week 2,
  Plasma levels concentrations
• Changes in plasma levels of calcineurin & mTOR inhibitors | Week 12,
  Plasma levels concentrations
• Changes in plasma levels of calcineurin & mTOR inhibitors | Week 24,
  Plasma levels concentrations
• Changes in plasma levels of calcineurin & mTOR inhibitors | Week 48
  Plasma levels concentrations
• B/F/TAF plasma levels | Week 4
  B/F/TAF PK
• Change in mGFR (iohexol clearance) | Baseline,
  evolution of mGFR
• Change in mGFR (iohexol clearance) | Week 48
  evolution of mGFR
• Change in bone markers | Baseline,
  bone markers and bone mineral density evolution
• Change in bone mineral density | Baseline,
  bone markers and bone mineral density evolution
• Change in bone mineral density | Week 48
  bone markers and bone mineral density evolution
• Change in bone markers | Week 48
  bone markers and bone mineral density evolution
• Incidence of proximal tubulopathy | W48
  (hypouricemia, hypophosphatemia, low molecular weight proteinuria, orthoglycemic glycosuria) analysis
• Incidence of proximal tubulopathy | Baseline
  (hypouricemia, hypophosphatemia, low molecular weight proteinuria, orthoglycemic glycosuria) analysis
• Change in eGFR evaluated with plasma or serum Cystatin C | Baseline
  evolution of eGFR
• Change in eGFR evaluated with plasma or serum Cystatin C | Week 48
  evolution of eGFR
• graft Survival | Baseline to Week 48
  defined as the necessity to return to dialysis, or death
• Change in plasma metabolome | Baseline to Week 48
  (Indoxyl sulfate, indole-3-acetic acid, Hippuric acid, para-cresol sulfate, 3-carboxy-4-methyl-5-propyl-2-furanpropanoic acid (CMPF) analysis
• Incidence of Grade ≥3 adverse events up | baseline to Week48
  adverse event≥3 reported
• Incidence of specific calcineurin inhibitors | Baseline to Week 48
  histological renal damage performed (if graft biopsy )
• Antiretroviral therapy changes during the follow-up through | Baseline to Week 48
  Antiretroviral therapy changes
• Calcineurin & mTOR inhibitors' drug dose changes | Baseline to Week 48
  Calcineurin & mTOR inhibitors' drug dose changes
• Proportion of patients with plasma HIV RNA ≤ 50 cp/mL | Week 48
  Proportion of patients with plasma HIV RNA ≤ 50 cp/mL
• Change CD4 cell count, ratio CD4/CD8 | Baseline
  Immunology evolution
• Change CD4 cell count, ratio CD4/CD8 | Week 24
  Immunology evolution
• Change CD4 cell count, ratio CD4/CD8 | Week 48
  Immunology evolution
• proportion of participants with virological failure | Baseline to Week 48
  defined as two consecutive HIV RNA VL>50 copies/mL or a HIV RNA >50 copies/mL followed by a study treatment discontinuation"
• Change in GSS* after switch to B/F/TAF Genotypic Susceptibility Score (GSS) to B/F/TAF | baseline to Week 48
  GSS ≥ 2
• Adherence, HIV Treatment Satisfaction | Baseline,
  adherence and satisfactory questionnaire
• Adherence, HIV Treatment Satisfaction | Week12,
  adherence and satisfactory questionnaire
• Adherence, HIV Treatment Satisfaction | ,Week 24,
  adherence and satisfactory questionnaire
• Adherence, HIV Treatment Satisfaction | Week36,
  adherence and satisfactory questionnaire
• Adherence, HIV Treatment Satisfaction | Week48
  adherence and satisfactory questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Henri Mondor, Créteil
  - Hopital Hotel Dieu, Nantes